CLINICAL TRIAL: NCT02860169
Title: Effects of Cold and/or Flu on Motivation, Mood and Cognitive Performance in Otherwise Healthy Individuals
Brief Title: Motivation, Brain Function and Mood in Individuals With Cold and/or Flu
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to GSK concerns that the data collected in this study could not support reliable interpretation of assessments and conclusions on the primary objectives.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 205689
Record Dates: First submitted 2016-06-28; First posted 2016-08-09 (Estimated); Results first posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2018-01

CONDITIONS: Cognition
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Participants with cold and flu (Experimental): Eligible participants with cold and flu were instructed to answer the self administered questionnaire and participate in the assessment that included Picture Rating, Picture Surfing Task, Questionnaire and VAS scales, Cognitive Function Assessment, RTI, AST, ERT , RVP
  Interventions: Behavioral: Participants self-administered questionnaire and assessment
- Healthy participants (Placebo Comparator): Eligible healthy participants were instructed to answer the self administered questionnaire and participate in the assessment that included Picture Rating, Picture Surfing Task, Questionnaire and VAS scales, Cognitive Function Assessment, RTI, AST, ERT , RVP
  Interventions: Behavioral: Participants self-administered questionnaire and assessment

INTERVENTIONS:
Behavioral: Participants self-administered questionnaire and assessment — Participants self-administered questionnaire and assessment includes Picture Rating, Picture Surfing Task, Questionnaire and VAS scales, Cognitive Function Assessment, RTI, AST, ERT , RVP.

SUMMARY:
This study aim to adapt and test a novel indication of motivation in participants with cold & flu using the Picture Surfing Task (PST). The purpose of this task, in both healthy participants and those with cold & flu, will be to provide a measure of: 1) change in general motivation, 2) change in cold and flu-specific motivation, and 3) any change in general tendency to exert force to serve as a control.

DETAILED DESCRIPTION:
The study is designed in three parts. The first, Part A, is an online survey to select salient images (cold & flu related) to be used in the motivation task under investigation in Parts B and C. Part B is a pilot investigation of a novel measure of motivation, using a grip force cognitive task (PST, previously used in obesity literature) in a small group of participants with cold and flu compared to a group without. The result of this pilot study will inform task content and sample size for Part C. The final part will investigate the effects of cold and flu on motivation (using the PST), cognitive performance (using the Cambridge Cognition Cognitive Assessments [CANTAB] testing battery) and subjective mood and motivation in participants suffering from C&F and healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Part A: Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary informed consent confirmed online before completing the online survey.
* Part B and C: Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged between 18 and 65 years inclusive.
* Participant is male or female.
* Part A: Healthy adult with no chronic illness and currently free from acute illness.
* Part B and C: Good general and mental health with, in the opinion of the Investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history. Healthy group: Healthy adult with no chronic illness. Currently free from acute illness.

Exclusion Criteria:

* Woman who are known to be pregnant or who are intending to become pregnant over the duration of the study or who are breast-feeding.
* Parts B and C: Current (within 14 days of the start of the study) or regular use of any prescription, OTC and herbal medicine unless it will not interfere with study endpoints as determined by the principal investigator. Vitamin supplements and occasional doses of OTC paracetamol for pain relief/ treatment of cold and flu symptoms are permitted (with the exception of > 24 hours before study visits).
* Current or in the 30 days prior to dosing use of any drug known to induce or inhibit hepatic drug metabolism (e.g. barbiturates, theophylline, cimetidine, or erythromycin).
* Current or past use (within 2 years) if antidepressants or other psychoactive medication.
* Use of over the counter (OTC) analgesics/cold and flu treatments 24 hours prior to assessment visits in all parts of the study.
* Participant is colour blind.
* Recent history (within the last 5 years) of alcohol or other substance abuse.
* Participant must not be regular smokers (as defined - more than 3 per day or equivalent for e-cigarettes, chewing tobacco or pipes).
* Participant must not consume greater than 21 units of alcohol per week (male) and 14 units per week (female).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2016-11-24 (Actual); Study Completion 2016-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Brentford, Middlesex, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center at United Kingdom (UK).
Pre-assignment Details: This study was divided in 3 parts (A, B and C). Part A was an online survey, Parts B and C. Participants recruited separately for each part of the study based on the inclusion and exclusion criteria of respective part of the study. (46 [part A] + 20 [part B] + 48 [part C] = 114 enrolled in the study)
Groups:
- Overall Participants: The study consisted of three parts A (includes only healthy participants), B and C (both B and C included healthy and cold and flu participants). Recruitment is done separately for each part of the study, based on the inclusion and exclusion criteria set for the respective part of the study.
Period: Part A
Arm/Group | Overall Participants
Started (Part A recruited healthy participants for an online survey.) | 46
Healthy Participants | 46
Participants With Cold and Flu | 0
Completed | 35
Not Completed | 11
Not completed — Withdrawal by Subject | 1
Not completed — Other (Screening failure) | 6
Not completed — Other (Survey not completed) | 3
Not completed — Other (did not completed consent) | 1
Period: Part B
Arm/Group | Overall Participants
Started (Part B separately recruited healthy (control) and cold and flu participants.) | 20
Healthy Participants | 10
Participants With Cold and Flu | 10
Completed | 9
Not Completed | 11
Not completed — Other (Screening failure) | 10
Not completed — Withdrawal by Subject | 1
Period: Part C
Arm/Group | Overall Participants
Started (Part C separately recruited healthy (control) and cold and flu participants.) | 48
Healthy Participants | 6
Participants With Cold and Flu | 42
Completed | 47
Not Completed | 1
Not completed — Other (Screening failure) | 1

BASELINE CHARACTERISTICS:
Population: All the participants who participated in any part of the study (part A, B or C).
Groups:
- Healthy Participants: Eligible healthy participants were instructed to answer the self administered questionnaire and participate in the assessment that included Picture Rating, Picture Surfing Task, Questionnaire and visual analogue scale (VAS), Cognitive Function Assessment, Reaction time (RTI), Attention switching task (AST), Emotional recognition task (ERT) , Rapid visual information processing (RVP).
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | Participants With Cold and Flu | Total
Number analyzed (Participants) | 62 | 52 | 114
Age, Customized [Mean (Standard Deviation); unit: Years]
  Mean Age | 34.38 (11.01) | 31.3 (10.98) | 32.91 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 25 | 60
  Male | 27 | 27 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 28 | 42
  Asian | 1 | 18 | 19
  Mixed | 0 | 1 | 1
  Arab | 0 | 1 | 1
  Black | 4 | 1 | 5
  Not collected (Part A participants) | 46 | 0 | 46

OUTCOME MEASURES:

1. Primary Outcome: Liking Rating on 11 Point Likert Scale (0-10 - 0 = Not at All; 10 = Like Extremely)
Description: Participants will be asked to rate a selection of images relevant to cold and flu on an 11 point Likert scale of "how much do you like this image?" from 0 = "Not at all" to 10 = "Extremely like" (In Part A of the study).
Time Frame: At Screening
Population: No participant data were analysed for the study as it was terminated due to concerns relating to procedures for data collection. Based on these concerns, GlaxoSmithKline (GSK) is not confident that the data collected in this study could support reliable interpretation of the assessments and conclusions on the primary objectives of the study.
Arm/Group | Participants With Cold and Flu | Healthy Participants
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Reaction Time (RTI) Milliseconds (ms) From the Reaction Time Task in Participants Suffering From Cold and Flu Versus Healthy Participants
Description: Change in RTI will be measured by the five-choice reaction time task. The participant will hold down a button at the bottom of the screen until a yellow spot appears in one of the five circles at the top of the screen. Median from five-choice reaction time (the median duration between the onset of the stimulus and the release of the button) will be measured (In Part B of the study).
Time Frame: Day 1
Population: No participant data were analysed for the study as it was terminated due to concerns relating to procedures for data collection. Based on these concerns, GSK is not confident that the data collected in this study could support reliable interpretation of the assessments and conclusions on the primary objectives of the study.
Arm/Group | Participants With Cold and Flu | Healthy Participants
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change in Emotional Recognition Task (ERT) Score (Number of Total Hits) in Participants Suffering From Cold and Flu Versus Healthy Participants
Description: Change in ERT will be measured by displaying Morphed images of real participant's facial features, each showing a specific emotion on the screen for 200ms. The participant will need to decide from 6 options which emotion the face is displaying. Change in ERT (total hits) which is calculated from the number of problems during assessment blocks, on which the participant chose the correct emotion (In Part B of the study).
Time Frame: Day 1
Population: as for outcome 2
Arm/Group | Participants With Cold and Flu | Healthy Participants
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Change in Rapid Visual Information Processing (RVP) A Prime (RVP A') in Participants Suffering From Cold and Flu Versus Healthy Participants
Description: RVP A Prime will be measured with the help of a white box appears in the centre of computer screen inside which digits, from 2 to 9, appear in a pseudo-random order, at the rate of 100 digits per minute. Participants are requested to detect target sequences of digits (for example, 2-4-6, 3-5-7, 4-6-8) and to register responses using the press pad. RVP A Prime is the signal detection measure of sensitivity to the target, regardless of response tendency (the expected range is 0.00 to 1.00; bad to good). In essence, this metric is a measure of how good the participant is at detecting target sequences (In Part B of the study).
Time Frame: Day 1
Population: as for outcome 2
Arm/Group | Participants With Cold and Flu | Healthy Participants
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Change in Attention Switching Task (AST) Score (Congruency Cost [ms]) in Participants Suffering From Cold and Flu Versus Healthy Participants
Description: Change in AST score is a measure of executive attention. The test displays an arrow which can appear on either side of the screen (right or left) and can point in either direction (to the right or to the left). Each trial displays a cue at the top of the screen that indicates to the participant whether they have to press the right or left button according to the "side on which the arrow appeared" or the "direction in which the arrow was pointing". AST congruency cost (median; ms) will be measured as the difference between the median latency of response (from stimulus appearance to button press) on the trials that were congruent versus the trials that were incongruent. Calculated by subtracting the median congruent latency (ms) from the median incongruent latency. Close to zero: less variation in latencies across congruent and incongruent trials. A positive score: participant is faster on congruent trials and a negative score: participant is faster on incongruent trials (in Part C).
Time Frame: Day 1
Population: as for outcome 2
Arm/Group | Participants With Cold and Flu | Healthy Participants
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Change in Mood and Motivation Visual Analogue Scale (VAS) Change (Millimeter[mm]) in Participants Suffering From Cold and Flu Versus Healthy Participants
Description: VAS of 100mm line will be used to assess subjective ratings of mood and motivation. For mood participants will be asked to rate their current mood under the headings of alertness, pleasure/displeasure and anxiety. Motivation will be assessed by asking participants to rate their current motivation under six different headings e.g. general motivation, motivation to engage with friends and family and motivation to perform leisure activities (In Part B of the study).
Time Frame: Day 1
Population: as for outcome 2
Arm/Group | Participants With Cold and Flu | Healthy Participants
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: No participant data was analyzed for adverse events in this study as it was terminated early due to concerns relating to procedures for data collection, handling, and transfer that potentially impacted the integrity of the study data.
Arm/Group | Participants With Cold and Flu | Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study was terminated due to GSK concerns that the data collected in this study could not support reliable interpretation of the assessments and conclusions on the primary objectives of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.